CLINICAL TRIAL: NCT07362329
Title: Use of Resistive Exercise Snacks to Improve Upper Body Fitness in Graduate Students
Brief Title: Use of Exercise Snacks to Improve Upper Body Fitness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Alexander Rothstein, Assistant Professor, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NYIT IRB-2026-396 Title:
Record Dates: First submitted 2026-01-06; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Muscle Strength; Muscle Power; Physical Endurance
Keywords: Exercise snacks; resistance exercise; upper body fitness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A submaximal repeated effort exercise snack (SMR_ES) (Experimental): The SMR_ES group will perform approximately 33% of their individual number of maximal push-up and maximal plank time, three times per day, three days per week.
  Interventions: Behavioral: Submaximal Repeated Exercise Snack
- A maximal effort one-time exercise snack (MO_ES) (Experimental): The MO_ES group will perform the maximal number of push-ups and hold a plank position for their maximal time, once per day, three days per week.
  Interventions: Behavioral: Maximal One-Time Exercise Snack
- Control group (No Intervention): Continues usual activity with no upper body resistive exercise.

INTERVENTIONS:
Behavioral: Submaximal Repeated Exercise Snack — Participants perform frequent, low-dose submaximal upper-body exercise snacks spread throughout the day. The SMR_ES group will perform approximately 33% of their individual number of maximal push-up and maximal plank time, three times per day, three days per week.
  Arms: A submaximal repeated effort exercise snack (SMR_ES)
Behavioral: Maximal One-Time Exercise Snack — Participants perform a single daily maximal-effort upper-body exercise snack. The MO_ES group will perform the maximal number of push-ups and hold a plank position for their maximal time, once per day, three days per week.
  Arms: A maximal effort one-time exercise snack (MO_ES)

SUMMARY:
This study will examine the effects of an upper-body resistance "exercise snack" (ES) protocol on upper-body strength, endurance, and power. Participants will be randomly assigned to one of three groups: a submaximal effort repeated throughout the exercise day ES group, a maximal effort performed once per exercise day ES group, and a control group that continues usual activity (Control: no resistance exercise). Both exercise groups will perform two exercises, push-ups and planks, three days per week. The submaximal repeated effort ES group (SMR_ES) will perform approximately 33% of the maximal number of push-ups and maintain a plank position for 33% of maximal time, three times per day. The maximal once-per-day effort ES group (MO_ES) will perform the maximal number of push-ups and maintain a plank position for maximal time, once per day. Therefore, both ES groups (SMR_ES and MO_ES) will perform the same weekly volume (repetitions and time) of both exercises across the six-week intervention period.

Before and after the six-week intervention period, all participants will undergo testing to assess upper-body performance. Outcome measures will include push-up endurance (maximum repetitions), plank endurance (maximum time), push-up power (assessed using force plates), and maximal push strength (assessed using hand-held dynamometry). Pre- and post-intervention changes in outcomes will be compared among all three groups. If significant changes are identified, additional comparisons will be conducted between the SMR_ES and Control groups, as well as between the SMR_ES and MO_ES groups.

The primary aim of this study is to determine whether repeated submaximal efforts performed three times per day, three days per week, increase upper-body endurance, power, and strength compared to a control group performing no resistance exercise. The secondary aim is to determine whether submaximal efforts performed three times per day, three days per week, produce changes in upper-body strength, endurance, and power that are not different from maximal efforts performed once per day, three days per week. These aims address whether exercise distribution influences strength and power adaptations beyond total weekly volume. The findings may help inform time-efficient, lower subjective-effort resistance training strategies that can be implemented in educational, athletic, or general fitness settings.

DETAILED DESCRIPTION:
The academic demands imposed on graduate students present a barrier to performing regular resistive exercise and promote a sedentary lifestyle, which can lead to losses in upper-body strength, power, and endurance.

There are many causes of loss of lean body mass (LBM) in the general population. Decreases in strength and LBM typically begin between thirty and forty years of age and progress at a rate of 3-10% per decade. After the age of 70, the rate of LBM loss and strength decline accelerates to approximately 3% per year. These changes may be attributed to immobilization, loss of appetite, muscular dystrophies, chronic disease, aging, and sedentary behavior. By age 65, difficulty with dressing, transferring, walking, and toileting occurs at rates between 14% and 17%. By age 75, the incidence of difficulty increases to between 20% and 27%, and by age 85, difficulty with dressing, bathing, walking, toileting, and transferring increases to between 26% and 36%. Decreases in LBM and strength are strong indicators of negative health outcomes and represent one of the primary contributors to sarcopenia, alongside anorexia, dehydration, and cachexia. Loss of LBM combined with obesity further increases the risk of developing type II diabetes due to the role of skeletal muscle in glycemic control. Reductions in LBM also negatively affect bone density and metabolic rate.

Resistance training is one of the most effective interventions for improving physical performance and long-term health across the lifespan. Resistance training enhances muscular strength, endurance, and neuromuscular control, all of which are essential for optimal movement, joint stability, and performance of daily functional activities. Resistance exercise stimulates muscle hypertrophy, improves motor unit recruitment, increases LBM, and supports metabolic health through improved insulin sensitivity and elevated resting metabolic rate.

In older adults, resistance training increases muscle mass, strength, and power, while reducing difficulty performing daily activities and supporting independence with aging. Moderate-intensity, short-term resistance training significantly improves insulin sensitivity and HbA1c levels in older adults. In older women, resistance training reduces age-related declines in cortical bone health and bone mineral density of the hip and spine. Resistance training also reduces mild to severe depressive symptoms, thereby improving quality of life across age groups.

The American College of Sports Medicine (ACSM), American Heart Association (AHA), National Institutes of Health (NIH), and National Health Service (NHS) recommend performing resistance exercises at least twice per week for all major muscle groups, including the legs, hips, back, chest, abdomen, shoulders, and arms. These exercises are generally recommended at moderate intensity, characterized by muscular fatigue after completing 12-15 repetitions.

Despite the known benefits of resistance exercise, many individuals face barriers to consistent participation. Physical limitations associated with aging, chronic health conditions, psychological factors (e.g., lack of motivation, fear of injury, embarrassment), limited transportation, financial constraints, and environmental factors such as weather can all negatively affect adherence.

Among graduate students, time constraints related to academic workload are a primary barrier to regular resistance exercise and promote sedentary behavior. Previous studies have demonstrated declines in fitness and exercise participation during graduate training. Limited institutional support for physical activity and financial constraints further exacerbate barriers to consistent resistance training.

A potential solution to declining fitness among graduate students is the integration of resistive "exercise snacks" (ES). Exercise snacks are brief bouts of exercise lasting 1-5 minutes, separated by short rest periods, and performed multiple times per day. These sessions can be completed as little as three times per week.

Current literature strongly supports the viability of the ES approach. A 2024 systematic review by Yin et al. examining 11 randomized controlled trials found that ES protocols improved strength, flexibility, and balance in older adults without requiring equipment, while reducing common barriers such as time constraints and access limitations. Additional randomized trials have demonstrated improvements in cardiorespiratory fitness, muscular strength, power, and adherence using minimal-volume ES protocols across diverse populations.

Collectively, the literature supports ES as a time-efficient and effective training strategy for improving muscular and cardiovascular outcomes while enhancing adherence among populations facing barriers to traditional exercise. However, research examining upper-body resistance-based ES in young adult populations remains limited.

The objective of this study is to determine the effects of a six-week upper-body ES program performed at submaximal intensities on upper-body strength, power, endurance, participant retention, adherence, and satisfaction. The study aims to determine whether short-duration, repeated submaximal ES performed multiple times per day, three days per week, elicits positive adaptations in upper-body muscular performance among graduate students who do not regularly engage in resistance training.

It is hypothesized that the ES group will demonstrate greater improvements in upper-body strength and endurance compared to a control group maintaining usual physical activity. A secondary hypothesis is that outcomes in the ES group will not differ from those observed in a maximal-intensity, once-daily resistance exercise group performing the same exercises three days per week. A third hypothesis is that the ES group will demonstrate greater participant retention, adherence, and satisfaction compared to the maximal-intensity exercise group.

Investigating the effects of upper-body resistive ES on muscular performance in graduate students may identify an accessible, time-efficient, and lower-effort training strategy capable of improving strength, power, and adherence despite substantial academic demands.

ELIGIBILITY:
Inclusion Criteria

Healthy, as determined by self-reported health history

Enrolled as a college or university student (full-time or part-time)

Not currently participating in a structured upper-body resistance training program

No participation in upper-body resistance training (e.g., weightlifting, calisthenics, CrossFit, bodyweight strength programs) for ≥ 3 months prior to study enrollment

Willing and able to perform maximal and submaximal push-up and plank exercises

Willing to refrain from initiating any new upper-body resistance training during the study period

Able to provide written informed consent

Exclusion Criteria

Current participation in an upper-body resistance training program or engagement in upper-body strength training within the past 3 months

History of upper extremity, shoulder, elbow, wrist, or trunk injury within the past 6 months that could limit exercise performance

History of neurological, cardiovascular, metabolic, or musculoskeletal disorders that contraindicate resistance exercise

Current pain or discomfort in the shoulders, elbows, wrists, hands, neck, or low back during pushing or plank activities

Previous surgery to the upper extremities or spine within the past 12 months

Use of medications that may significantly affect muscle performance, fatigue, or neuromuscular function

Pregnancy or suspected pregnancy

Any condition deemed by the investigators to pose an increased risk during maximal or repeated resistance exercise

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Upper Body Push Strength | Change from baseline after 6 weeks
  Upper-body muscular strength will be assessed using a hand-held dynamometer during a standardized pushing task. Participants will push a barbell upward against an immovable strap connected to a pull dynamometer. Peak force output (Newtons) will be recorded.
Push-Up Endurance (Repetitions) | Change from baseline after 6 weeks.
  Upper-body muscular endurance will be assessed by the maximum number of push-ups completed using standardized form criteria.
Plank Endurance (Seconds) | Change from baseline after 6 weeks
  Core and upper-body endurance will be assessed by the maximum duration (seconds) participants can maintain a standardized plank position.

SECONDARY OUTCOMES:
Upper-Body Power - Peak Force (Newtons) | Change from baseline after 6 weeks.
  Upper-body power will be assessed during maximal push-up efforts performed on force plates. Peak force output (Newtons) will be recorded.
Upper-Body Power - Time to Task Completion (Seconds) | Change from baseline after 6 weeks
  Time to completion (seconds) of maximal push-up efforts performed on force plates will be recorded as an additional indicator of power output.

OTHER OUTCOMES:
Upper-Body Power - Mean Force (Newtons) | Observed over 6 weeks.
  Mean force output (Newtons) during maximal push-up efforts performed on force plates will be recorded.
Participant Retention (%) | Observed over 6 weeks
  Participant retention will be calculated as the percentage of enrolled participants who complete the full 6-week intervention.
Protocol Adherence (%) | Observed over 6 weeks
  Adherence to the exercise protocol will be assessed as the percentage of supervised exercise sessions completed relative to the total number prescribed.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Rothstein, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We will upload our shared anonymized data using DryAd.
Supporting Information: Study Protocol, SAP
Time Frame: The information will be available May 2026 and remain for 5 years.
Access Criteria: Access will require access to DryAd or a request for access to the researchers.

REFERENCES:
- [Background] Marijancic V, Grubic Kezele T, Peharec S, Dragas-Zubalj N, Pavicic Zezelj S, Starcevic-Klasan G. Relationship between Physical Activity and Sedentary Behavior, Spinal Curvatures, Endurance and Balance of the Trunk Muscles-Extended Physical Health Analysis in Young Adults. Int J Environ Res Public Health. 2023 Oct 18;20(20):6938. doi: 10.3390/ijerph20206938. PMID 37887676
- [Background] Jett KM, Daniels BT, Brigance M, Passarelli JL, Howie EK. A Qualitative Description of Graduate Students' Perceived Decline in Physical Activity from Undergraduate School. Int J Exerc Sci. 2024 Aug 1;17(5):1038-1055. doi: 10.70252/ORGX1052. eCollection 2024. PMID 39257547
- [Background] Stork MJ, Marcotte-Chenard A, Jung ME, Little JP. Exercise in the workplace: examining the receptivity of practical and time-efficient stair-climbing "exercise snacks". Appl Physiol Nutr Metab. 2024 Jan 1;49(1):30-40. doi: 10.1139/apnm-2023-0128. Epub 2023 Sep 25. PMID 37748202
- [Background] DiFrancisco-Donoghue J, Werner W, Douris PC. Comparison of once-weekly and twice-weekly strength training in older adults. Br J Sports Med. 2007 Jan;41(1):19-22. doi: 10.1136/bjsm.2006.029330. Epub 2006 Oct 24. PMID 17062657
- [Background] Brandt T, Schwandner CTL, Schmidt A. Resistance exercise snacks improve muscle mass in female university employees: a prospective, controlled, intervention pilot-study. Front Public Health. 2024 Feb 6;12:1347825. doi: 10.3389/fpubh.2024.1347825. eCollection 2024. PMID 38379679
- [Background] Perkin OJ, McGuigan PM, Stokes KA. Exercise Snacking to Improve Muscle Function in Healthy Older Adults: A Pilot Study. J Aging Res. 2019 Oct 3;2019:7516939. doi: 10.1155/2019/7516939. eCollection 2019. PMID 31687210
- [Background] Yin M, Zheng H, Bai M, Huang G, Chen Z, Deng S, Lyu M, Deng J, Zhang B, Li H, Zhang X, Liu Q, Little JP, Li Y. Effects of Integrating Stair Climbing-Based Exercise Snacks Into the Campus on Feasibility, Perceived Efficacy, and Participation Perspectives in Inactive Young Adults: A Randomized Mixed-Methods Pilot Study. Scand J Med Sci Sports. 2024 Dec;34(12):e14771. doi: 10.1111/sms.14771. PMID 39587826
- [Background] Yin M, Deng S, Chen Z, Zhang B, Zheng H, Bai M, Li H, Zhang X, Deng J, Liu Q, Little JP, Li Y. Exercise snacks are a time-efficient alternative to moderate-intensity continuous training for improving cardiorespiratory fitness but not maximal fat oxidation in inactive adults: a randomized controlled trial. Appl Physiol Nutr Metab. 2024 Jul 1;49(7):920-932. doi: 10.1139/apnm-2023-0593. Epub 2024 Apr 3. PMID 38569204
- [Background] Jenkins EM, Nairn LN, Skelly LE, Little JP, Gibala MJ. Do stair climbing exercise "snacks" improve cardiorespiratory fitness? Appl Physiol Nutr Metab. 2019 Jun;44(6):681-684. doi: 10.1139/apnm-2018-0675. Epub 2019 Jan 16. PMID 30649897
- [Background] Wang T, Laher I, Li S. Exercise snacks and physical fitness in sedentary populations. Sports Med Health Sci. 2024 Feb 27;7(1):1-7. doi: 10.1016/j.smhs.2024.02.006. eCollection 2025 Jan. PMID 39649791
- [Background] Western MJ, Welsh T, Keen K, Bishop V, Perkin OJ. Exercise snacking to improve physical function in pre-frail older adult memory clinic patients: a 28-day pilot study. BMC Geriatr. 2023 Aug 4;23(1):471. doi: 10.1186/s12877-023-04169-6. PMID 37542234
- [Background] Rodriguez MA, Quintana-Cepedal M, Cheval B, Thogersen-Ntoumani C, Crespo I, Olmedillas H. Effect of exercise snacks on fitness and cardiometabolic health in physically inactive individuals: systematic review and meta-analysis. Br J Sports Med. 2026 Jan 19;60(2):133-141. doi: 10.1136/bjsports-2025-110027. PMID 41057224
- [Background] Hanson, Melanie. "Student Loan Debt Statistics" EducationData.org, 2025-08-08,
- [Background] Herazo-Beltran Y, Pinillos Y, Vidarte J, Crissien E, Suarez D, Garcia R. Predictors of perceived barriers to physical activity in the general adult population: a cross-sectional study. Braz J Phys Ther. 2017 Jan-Feb;21(1):44-50. doi: 10.1016/j.bjpt.2016.04.003. Epub 2017 Jan 14. PMID 28442074
- [Background] Scroggs GJ, Battista RA, Kappus RM. Bridging the Gap: Promoting Physical Activity in College-Aged Students. Prev Chronic Dis. 2025 Jul 10;22:E36. doi: 10.5888/pcd22.250118. No abstract available. PMID 40638806
- [Background] Douris PC, D'Agostino NA, Mathew SK, et al. The Physiological and Psychological Effects of the First Year of an Entry-Level Physical Therapist Education Program on Students. Journal of Physical Therapy Education. 2020;34(3):186-191
- [Background] Stephens MB, Cochran C, Hall JM, Olsen C. Physical fitness during medical school: a 4-year study at the Uniformed Services University. Fam Med. 2012 Nov-Dec;44(10):694-7. PMID 23148000
- [Background] Rimmer JH, Riley B, Wang E, Rauworth A, Jurkowski J. Physical activity participation among persons with disabilities: barriers and facilitators. Am J Prev Med. 2004 Jun;26(5):419-25. doi: 10.1016/j.amepre.2004.02.002. PMID 15165658
- [Background] Milner JD, DeFroda SF, Cruz AI Jr. Fitness habits and barriers to exercise during residency training. Orthop Rev (Pavia). 2020 Nov 24;12(3):8507. doi: 10.4081/or.2020.8507. eCollection 2020 Nov 24. PMID 33312484
- [Background] Gomez-Lopez M, Gallegos AG, Extremera AB. Perceived barriers by university students in the practice of physical activities. J Sports Sci Med. 2010 Sep 1;9(3):374-81. eCollection 2010. PMID 24149629
- [Background] Cottrell R, Girvan J, McKenzie J, Seabert D, Sterns P. Principles and Foundations of Health Promotion and Education. 7th ed. Pearson Education; 2018.
- [Background] Lindsay Smith G, Banting L, Eime R, O'Sullivan G, van Uffelen JGZ. The association between social support and physical activity in older adults: a systematic review. Int J Behav Nutr Phys Act. 2017 Apr 27;14(1):56. doi: 10.1186/s12966-017-0509-8. PMID 28449673
- [Background] NHS. Physical activity guidelines for adults aged 19 to 64. NHS. Published May 22, 2024.
- [Background] Physical Activity and Your Heart - Recommendations | NHLBI, NIH. www.nhlbi.nih.gov. Published March 24, 2022.
- [Background] American Heart Association. American Heart Association Recommendations for Physical Activity in Adults and Kids. American Heart Association. Published January 19, 2024
- [Background] American College of Sports Medicine. Physical Activity Guidelines. ACSM. Published 2025.
- [Background] Jiahao L, Jiajin L, Yifan L. Effects of resistance training on insulin sensitivity in the elderly: A meta-analysis of randomized controlled trials. J Exerc Sci Fit. 2021 Oct;19(4):241-251. doi: 10.1016/j.jesf.2021.08.002. Epub 2021 Aug 19. PMID 34552636
- [Background] Gordon BR, McDowell CP, Hallgren M, Meyer JD, Lyons M, Herring MP. Association of Efficacy of Resistance Exercise Training With Depressive Symptoms: Meta-analysis and Meta-regression Analysis of Randomized Clinical Trials. JAMA Psychiatry. 2018 Jun 1;75(6):566-576. doi: 10.1001/jamapsychiatry.2018.0572. PMID 29800984
- [Background] Massini DA, Nedog FH, de Oliveira TP, Almeida TAF, Santana CAA, Neiva CM, Macedo AG, Castro EA, Espada MC, Santos FJ, Pessoa Filho DM. The Effect of Resistance Training on Bone Mineral Density in Older Adults: A Systematic Review and Meta-Analysis. Healthcare (Basel). 2022 Jun 17;10(6):1129. doi: 10.3390/healthcare10061129. PMID 35742181
- [Background] Hong AR, Kim SW. Effects of Resistance Exercise on Bone Health. Endocrinol Metab (Seoul). 2018 Dec;33(4):435-444. doi: 10.3803/EnM.2018.33.4.435. PMID 30513557
- [Background] Liu CJ, Latham NK. Progressive resistance strength training for improving physical function in older adults. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD002759. doi: 10.1002/14651858.CD002759.pub2. PMID 19588334
- [Background] Hunter GR, McCarthy JP, Bamman MM. Effects of resistance training on older adults. Sports Med. 2004;34(5):329-48. doi: 10.2165/00007256-200434050-00005. PMID 15107011
- [Background] Al-Ozairi E, Alsaeed D, Alroudhan D, Voase N, Hasan A, Gill JMR, Sattar N, Welsh P, Gray CM, Boonpor J, Celis-Morales C, Gray SR. Skeletal Muscle and Metabolic Health: How Do We Increase Muscle Mass and Function in People with Type 2 Diabetes? J Clin Endocrinol Metab. 2021 Jan 23;106(2):309-317. doi: 10.1210/clinem/dgaa835. PMID 33336682
- [Background] Jun JE, Lee SE, Lee YB, Kim G, Jin SM, Jee JH, Kim JH. Low Skeletal Muscle Mass Accompanied by Abdominal Obesity Additively Increases the Risk of Incident Type 2 Diabetes. J Clin Endocrinol Metab. 2023 Apr 13;108(5):1173-1180. doi: 10.1210/clinem/dgac662. PMID 36394524
- [Background] von Haehling S, Morley JE, Anker SD. An overview of sarcopenia: facts and numbers on prevalence and clinical impact. J Cachexia Sarcopenia Muscle. 2010 Dec;1(2):129-133. doi: 10.1007/s13539-010-0014-2. Epub 2010 Dec 17. PMID 21475695
- [Background] Falls and Fractures in Older Adults: Causes and Prevention. National Institute on Aging. Accessed November 20, 2025.
- [Background] Landi F, Calvani R, Martone AM, Salini S, Zazzara MB, Candeloro M, Coelho-Junior HJ, Tosato M, Picca A, Marzetti E. Normative values of muscle strength across ages in a 'real world' population: results from the longevity check-up 7+ project. J Cachexia Sarcopenia Muscle. 2020 Dec;11(6):1562-1569. doi: 10.1002/jcsm.12610. Epub 2020 Nov 4. PMID 33147374
- [Background] Brown RT, Diaz-Ramirez LG, Boscardin WJ, Cappola AR, Lee SJ, Steinman MA. Changes in the Hierarchy of Functional Impairment From Middle Age to Older Age. J Gerontol A Biol Sci Med Sci. 2022 Aug 12;77(8):1577-1584. doi: 10.1093/gerona/glab250. PMID 34498040
- [Background] Drescher C, Konishi M, Ebner N, Springer J. Loss of muscle mass: current developments in cachexia and sarcopenia focused on biomarkers and treatment. J Cachexia Sarcopenia Muscle. 2015 Dec;6(4):303-11. doi: 10.1002/jcsm.12082. Epub 2015 Nov 18. PMID 26676067
- [Background] Leon AS. Attenuation of Adverse Effects of Aging on Skeletal Muscle by Regular Exercise and Nutritional Support. Am J Lifestyle Med. 2016 Jun 23;11(1):4-16. doi: 10.1177/1559827615589319. eCollection 2017 Jan-Feb. PMID 30202306
- [Background] Volpi E, Nazemi R, Fujita S. Muscle tissue changes with aging. Curr Opin Clin Nutr Metab Care. 2004 Jul;7(4):405-10. doi: 10.1097/01.mco.0000134362.76653.b2. PMID 15192443
- [Background] Keller K, Engelhardt M. Strength and muscle mass loss with aging process. Age and strength loss. Muscles Ligaments Tendons J. 2014 Feb 24;3(4):346-50. eCollection 2013 Oct. PMID 24596700